CLINICAL TRIAL: NCT06495606
Title: The Voice of Reflux: Typical Vocal Biomarkers in Patients With Gastroesophageal Reflux Disease
Brief Title: "The Voice of Reflux" - Backflow of Gastric Juice Leads to Irritation of the Vocal Folds: Are There Typical Differences in the Voice?
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-02361
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: GERD Gastroesophageal Reflux Disease; Laryngopharyngeal Reflux Disease
Keywords: GERD; LPRD; Reflux; Voice; Vocal Biomarker
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GERD-Group: Patients with confirmed gastroesophageal reflux in diagnostics
  Interventions: Diagnostic Test: Voice sample; Recording with microphone + Questionnaire
- Non-GERD-Group: Patients with confirmed absence of gastroesophageal reflux in diagnostics
  Interventions: Diagnostic Test: Voice sample; Recording with microphone + Questionnaire

INTERVENTIONS:
Diagnostic Test: Voice sample; Recording with microphone + Questionnaire — Voice sample recording with microphone; afterwards digitalization and comparison between GERD and Non-GERD Group and also between GERD-Group before and after GERD treatment; searching for vocal biomarkers typical for GERD

SUMMARY:
If gastric juice refluxes back into the oesophagus and up into the throat/pharynx/mouth area, causing discomfort or injury, this is known as reflux disease (reflux). Classic symptoms include a burning pain in the middle of the upper abdomen, chest or throat (so-called heartburn), regurgitation of food (acid regurgitation), foreign body sensation in the throat area. There are also changes in the voice, hoarseness, difficulty clearing the throat, difficulty swallowing or a dry, irritating cough due to the chemical irritation of the vocal folds by the gastric juice. There are various causes of reflux. Often there is a weakness of the lower oesophageal sphincter or a hiatal hernia, which favours the reflux of gastric juice. Sometimes there are also movement disorders in the oesophagus or stomach with insufficiently efficient transport of food and liquids.

After a consultation with a specialist, three further standard examinations are ordered as a matter of priority for a proper reflux diagnosis:

* Gastroscopy: a tube-shaped camera can be used to view the mouth, pharynx, throat, oesophagus, stomach and the beginning of the duodenum and, if necessary, small tissue samples can be taken.
* Oesophageal manometry: A pressure measurement of the oesophagus can detect movement disorders or a malfunction of the oesophagus and sphincter.
* 24-hour impedance pH measurement: A small tube is placed in the oesophagus through the nose and left there for 24 hours. The probe measures how often gastric juice flows back to a certain level and how acidic this juice is.

These examinations allow reflux to be definitively diagnosed, possible causes to be identified, any further investigations to be considered and the best possible treatment to be suggested.

In these times of rapidly advancing digitalisation and increasing technical possibilities, we ask ourselves the following: If reflux changes the voice - would it be possible to detect reflux disease with voice samples the other way round? Studies are already underway in several other medical fields that are successfully analysing voice and speech samples and looking for typical changes in the voice pattern for diseases.

Our theory: Alterations typical for reflux can be found in voice samples. In future, voice samples can be used as a harmless, simple and inexpensive initial assessment for reflux.

The questions of our research project are therefore:

1. Do patients with confirmed reflux have a typical pattern of changes in their voice?
2. Can these changes be reliably determined via voice analyses?
3. Could a simple voice sample become the first basic examination for reflux patients in the future?

Procedure and duration of the study:

This project will be conducted exclusively at the Inselspital Bern (monocentric = 1 hospital, national = 1 country). All persons who receive the above-mentioned standard examination for a reflux clarification are eligible for participation. The standard examination will either confirm or rule out reflux. For our research project, we want to investigate two situations:

1. firstly, as a baseline, we would like to examine the voices of 47 participants with confirmed reflux and compare them with the voices of 47 participants with confirmed absence of reflux disease.
2. secondly, we would like to check the voices of participants with confirmed reflux again 5 months after the start of treatment and compare them with their initial situation.

Participants will complete a questionnaire and provide a voice sample (short simple recording into a microphone). Participation in the research project does not require any additional hospital visits or consultation appointments and lasts a maximum of 5 months.

The voice samples are then digitised, analysed, evaluated and searched for typical patterns of change by us in collaboration with the CSEM Neuchâtel (Centre Suisse Électronique et de Microtechnique). CSEM is an internationally recognised Swiss technology innovation centre that will help us with the sophisticated evaluation of the voice analyses. As these are simple voice recordings into a microphone, there are no additional clarifications, interventions or risks involved in participating. Data will be stored in encrypted form in a SharePoint database in strict compliance with all data protection regulations and will only be used for the agreed research project. Results are expected in 2025.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* Informed consent
* Undergoing gastroesophageal reflux diagnostic according to the current standard
* Basic reading skills in German or English

Exclusion Criteria:

* Age below 18
* No basic reading skills in German or English
* Diseases with altered voice
* Laryngopharyngeal surgery or interventions in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We include patients undergoing GERD diagnostic with esophagogastroduodenoscopy plus biopsies, high-resolution manometry and 24-hour impedance-pH-metry, according to the todays standard in reflux diagnostics, in the Bauchzentrum of University Hospital Bern Inselspital. After this standardized examination, there will be patients with confirmed gastroesophageal reflux disease as well as patients with confirmed absence of a GERD. Out of these patients, we collect N=47 patients with confirmed gastroesophageal reflux disease (GERD-Group) and N=47 patients with confirmed absence of gastroesophageal reflux disease as a control group (Non-GERD-Group).
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Identify typical vocal biomarkers in the voice sample of patients with GERD | First acoustic voice recording at enrollement after finishing diagnostic measurements in GERD and Non-GERD Group; in GERD Group additional second acoustic voice recording 5 months after start treatment
  After digitizing the vocal samples and audio pre-processing, we will extract audio features and identify the most dominating and discriminating characteristics of the signal. The following audio features will be analyzed: 1)Acoustic measures: Variation of periodicity analyzing Jitter and Shimmer, Harmonics-to-Noise-Ratio, Fundamental frequency of voice FO, Amplitude Perturbation Quotient and Pitch Perturbation Quotient and 2) Spectral analysis using the Fast-Fourier Transformation FFT with further analysis using the Mel-Spectrogram. The analysed audio features and Mel-spectrograms will be compared between participants with GERD and participants without GERD at baseline as well as between participants with GERD before and after their treatment. We want to identify, if the pre-treatment GERD-patients show significantly more pathologic acoustic measures, Mel-spectrograms or a typical combination of abnormalities.

SECONDARY OUTCOMES:
To identify if there is a consistent correlation between vocal biomarkers and described symptoms of reflux | Comparrison vocal biomarkers in voice recordings and results of questionnaire at enrollment and in GERD-Group additionally 5 months after start treatment
  Do the vocal biomarkers correlate with the reflux-related symptoms reported in the questionnaires; Analysis of "GERD HRQL"- and "RSI"-Score
To identify if there is a consistent correlation between vocal biomarkers and described vocal symptoms | Comparisson of vocal biomarkers in voice recording and symptoms in questionnaire at enrollement and additionally in GERD-Group 5 months after start treatment
  Do the vocal biomarkers correlate with the voice-related symptoms reported in the questionnaires; Analysis of "VHI-10"- and "VRQoL"-Score

CONTACTS AND LOCATIONS:
Overall Officials: Yves Borbély, Dr. med., Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Universitätsspital Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available